CLINICAL TRIAL: NCT06988566
Title: Telemedical Monitoring and Treatment of COPD Patients Associated With General Practice (TEMOKAP)
Brief Title: Reduced COPD Related Utilization of Healthcare Services and Increased Social Activities by Patients Offered a 24/7 Accessible Telehealth Service Based on the Epital Care Model.
Acronym: TEMOKAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ECM Klinikken APS (Network)
Responsible Party: Principal Investigator, Klaus Phanareth, Principal Investigator, MD, Ph.D., ECM Klinikken APS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: F-24055647
Record Dates: First submitted 2025-05-16; First posted 2025-05-25 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator): The placebo group received the usual care provided by the GP and other health relevant stakeholders.
  Interventions: Other: Intervention Group
- Intervention group (Active Comparator): The intervention were connected to the ECM response and coordination centre (RCC) which provided the participants with 24/7/365 access to assistance from certified RCC staff who were supported by eDoctors. Patients self-tracking activities (saturation, pulse, lung function, temperature and report on increased sputum, coughing, and shortness of breath) were monitored dayly by the RCC whoom would contact them in the event of signs of deterioration. The RCC staff together with the participant would make informed decisions, via phone or video call, on how to best manage the change in condition guided by the previous measures evaluated with graphs, including plotted trends. If there was a need for medical treatment, a treatment plan was drawn up with fixed follow-ups and a course plan.
  Interventions: Other: Intervention Group

INTERVENTIONS:
Other: Intervention Group — The intervention were connected to the ECM response and coordination centre (RCC) which provided the participants with 24/7/365 access to assistance from certified RCC staff who were supported by eDoctors. Patients self-tracking activities (saturation, pulse, lung function, temperature and report on increased sputum, coughing, and shortness of breath) were monitored dayly by the RCC whoom would contact them in the event of signs of deterioration. The RCC staff together with the participant would make informed decisions, via phone or video call, on how to best manage the change in condition guided by the previous measures evaluated with graphs, including plotted trends. If there was a need for medical treatment, a treatment plan was drawn up with fixed follow-ups and a course plan.
  Other Names: ECM Intervention

SUMMARY:
The purpose of this study (The TEMOKAP study) is to investigate whether home-based treatment with telemedicine and support from healthcare professionals can prevent acute exacerbations of COPD and avoid acute hospital admissions, and whether this will improve the participant's health status and quality of life. In other words, the project seeks to document how life with COPD can be made better and safer for all COPD patients.

The project is a collaboration between the University of Copenhagen, alles Lægehus (everyone's medical practice), Epital Health A/S, and Apopro.dk and will be conducted as a scientific study.

DETAILED DESCRIPTION:
Why the TEMOKAP Study? The TEMOKAP study represents a new treatment method where, with the help of modern technology and telemedicine, we can offer examination and treatment in your own home if a medical issue or an acute exacerbation of your chronic illness should arise. In a time of Corona, as Denmark is experiencing, this principle is fully in line with the Danish Health Authority's recommendations to protect our chronic patients and reduce the risk of infection.

What are the benefits of participating?

* Direct and easy daily access to medical/healthcare professional help regarding your COPD
* The possibility of receiving treatment in the safe environment of your own home
* Free delivery of medication to your home address, so you don't have to go to the pharmacy yourself
* Reduced risk of infection with the Corona virus and other infectious diseases
* Prevention of exacerbations of your COPD and avoidance of hospital admissions
* Increased co-determination in your own treatment process
* Freedom and security to live better with a chronic illness How does it work? The TEMOKAP study works "proactively", meaning it reacts and acts "before the damage is done". This has become possible through the tele-tools that you will be provided with and use daily to take measurements from home. Your measurements are analyzed daily by mathematical models that can help the TEMOKAP study's doctors and nurses predict exacerbations, so they can initiate treatment much earlier than normal.

As a participant in the TEMOKAP study, in addition to your usual medication, you will have two types of "acute medication" (antibiotics and corticosteroids) readily available at home. This means that our doctors and nurses can initiate treatment immediately if an exacerbation should occur. You avoid a lot of hassle with getting prescriptions and picking up medication at the pharmacy - and most importantly, you save time and can start treatment quickly. TEMOKAP study, participant information (v3) 2 The TEMOKAP study also has a strong focus on your well-being and safety and therefore offers an open emergency line where you can get in touch with qualified healthcare professionals who are always ready if you need help or support in your daily life.

What does participation involve? Initially, you will undergo a clinical examination by a doctor or nurse from the TEMOKAP study with a special focus on your COPD. We will adjust your medication if necessary, and together we will make a plan for your wishes and goals for the future. You will then decide whether you wish to participate in the TEMOKAP study, and if you meet the necessary criteria for participation, you will need to sign a "Consent Form". Once signed, you will be randomly placed in either an "active group" or a "control group".

Active group As a participant in the "active group", you will be provided with an electronic screen (tablet) with a direct connection to the TEMOKAP study's doctors and nurses, as well as a spirometer and an oximeter. You will be trained in how to use the equipment to take your daily measurements and learn how to contact us if you need to.

Treatment, access to doctors and nurses, all technical equipment, and the delivery of medication are completely free for you. The only thing you have to pay for is your usual medication and the acute medication that you need to have readily available at home. The acute medication costs approximately DKK 50 after subsidy.

Electronic screen (tablet) Spirometer Oximeter Your participation in the TEMOKAP study will last for one year. At the start of the project, after 6 months, and at the end of the project, we will collect a series of health information about your health, which we will analyze to investigate how you have been and to compare with a "control group". This will take place a total of three times, through questionnaires and consultations that you will be invited to.

You will continue to be affiliated with alles LægeHus, so you can contact and visit your own doctor, just as you usually do, and if you are connected to a hospital outpatient clinic, this will also continue - as usual.

Control group As a participant in the "control group", you will continue your treatment as usual through alles LægeHus. At the start of the project, after 6 months, and at the end of the project after 1 year, you will be contacted by one of the TEMOKAP study's staff members who will collect a series of health information about your health to investigate and analyze how you have been. The results will be compared with the "Active group" to investigate the effect of the two treatments. This will take place a total of three times, through questionnaires and consultations that you will be invited to or called about.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥ 45 years
* diagnosed with COPD according to the criteria of the GOLD guideline
* a score of minimum three out of six points in cognitive screening test (The Clock Test + Three-Word Recall Memory Test)
* must have the ability to provide oral or written informed consent
* must have access to the internet in their own home
* must own a smartphone
* must be able to use simple functions in web browsers.

Exclusion Criteria:

* unstable heart disease
* poorly regulated diabetes
* diagnosed with psychiatric conditions who leads to mental impaired functions
* unable to communicate in oral and written Danish.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2020-09-04 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-09-02 (Actual)

PRIMARY OUTCOMES:
WHO-5 Well-Being Index and 1b: Contacts to healthcare services associated with COPD, 1c: The Readiness and Enablement Index for Health Technology (READHY) questionnaire | From enrollment to the end of treatment at 12 month
  Patient's mental well-being was assessed by the WHO-5 Well-Being Index. This is a validated questionnaire that examines patients' mental well-being and can also indicate anxiety, stress, and depression.
  1b: Patients' contacts to healthcare services associated with COPD included general practice (GP), out-of-offices services, outpatient clinics and hospital admissions at T0, T1 and T2 in both groups. Baseline information on hospital admissions was also examined retrospectively 12 months from the date of inclusion. Data are only self-reported but were verified by the clinical co-investigators with interviews to ensure that the COPD-related outcomes were accurate.
  1c: The Readiness and Enablement Index for Health Technology (READHY) allows for a more systematic assessment of patient readiness for health technology, which includes dimensions of self-management capabilities (including emotional distress), perceived support and digital health literacy. Together with socio-demographic
Patients' contacts to healthcare services associated with COPD | From enrollment to the end of treatment at 12 month
  Patients' contacts to healthcare services associated with COPD included general practice (GP), out-of-offices services, outpatient clinics and hospital admissions at T0, T1 and T2 in both groups. Baseline information on hospital admissions was also examined retrospectively 12 months from the date of inclusion. Data are only self-reported but were verified by the clinical co-investigators with interviews to ensure that the COPD-related outcomes were accurate.

SECONDARY OUTCOMES:
The Readiness and Enablement Index for Health Technology (READHY) | From enrollment to the end of treatment at 12 month
  The Readiness and Enablement Index for Health Technology (READHY) allows for a more systematic assessment of patient readiness for health technology, which includes dimensions of self-management capabilities (including emotional distress), perceived support and digital health literacy. Together with socio-demographic

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Phanareth, MD, Ph.D., Principal Investigator — ECM Klinikken APS
Locations (1):
- The ECM Clinic, Søborg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected throughout the trial
Supporting Information: Study Protocol

REFERENCES:
- [Background] Rossen S, Kayser L, Vibe-Petersen J, Ried-Larsen M, Christensen JF. Technology in exercise-based cancer rehabilitation: a cross-sectional study of receptiveness and readiness for e-Health utilization in Danish cancer rehabilitation. Acta Oncol. 2019 May;58(5):610-618. doi: 10.1080/0284186X.2018.1562213. Epub 2019 Jan 30. PMID 30698060
- [Background] Kayser L, Rossen S, Karnoe A, Elsworth G, Vibe-Petersen J, Christensen JF, Ried-Larsen M, Osborne RH. Development of the Multidimensional Readiness and Enablement Index for Health Technology (READHY) Tool to Measure Individuals' Health Technology Readiness: Initial Testing in a Cancer Rehabilitation Setting. J Med Internet Res. 2019 Feb 12;21(2):e10377. doi: 10.2196/10377. PMID 30747717
- [Background] Jakobsen AS, Laursen LC, Rydahl-Hansen S, Ostergaard B, Gerds TA, Emme C, Schou L, Phanareth K. Home-based telehealth hospitalization for exacerbation of chronic obstructive pulmonary disease: findings from "the virtual hospital" trial. Telemed J E Health. 2015 May;21(5):364-73. doi: 10.1089/tmj.2014.0098. Epub 2015 Feb 5. PMID 25654366
- [Background] Krag T, Jorgensen EH, Phanareth K, Kayser L. Experiences With In-Person and Virtual Health Care Services for People With Chronic Obstructive Pulmonary Disease: Qualitative Study. JMIR Rehabil Assist Technol. 2023 Aug 14;10:e43237. doi: 10.2196/43237. PMID 37578832
- [Background] Phanareth K, Dam AL, Hansen MABC, Lindskrog S, Vingtoft S, Kayser L. Revealing the Nature of Chronic Obstructive Pulmonary Disease Using Self-tracking and Analysis of Contact Patterns: Longitudinal Study. J Med Internet Res. 2021 Oct 19;23(10):e22567. doi: 10.2196/22567. PMID 34665151
- [Background] Phanareth K, Vingtoft S, Christensen AS, Nielsen JS, Svenstrup J, Berntsen GK, Newman SP, Kayser L. The Epital Care Model: A New Person-Centered Model of Technology-Enabled Integrated Care for People With Long Term Conditions. JMIR Res Protoc. 2017 Jan 16;6(1):e6. doi: 10.2196/resprot.6506. PMID 28093379
- [Derived] Phanareth K, Purreskov GT, Nielsen EF, Bentsen AT, Schou L, Newman S, Kayser L. Reduced Chronic Obstructive Pulmonary Disease-Related Utilization of Health Care Services and Increased Social Activities by Patients Offered a 24/7 Accessible Telehealth Service Based on the Epital Care Model: Pragmatic Modified Stepped Wedge Randomized Controlled Trial. J Med Internet Res. 2025 Oct 22;27:e65300. doi: 10.2196/65300. PMID 41125235